CLINICAL TRIAL: NCT00000717
Title: The Safety and Efficacy of Clindamycin and Primaquine in the Treatment of Mild - Moderate Pneumocystis Carinii Pneumonia in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 044; 11019 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Primaquine; Infusions, Intravenous; Drug Evaluation; Drug Therapy, Combination; Administration, Oral; Acquired Immunodeficiency Syndrome; Clindamycin
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Primaquine; Clindamycin

INTERVENTIONS:
Drug: Primaquine
Drug: Clindamycin

SUMMARY:
To determine the safety and effectiveness of clindamycin and primaquine in the treatment of mild Pneumocystis carinii pneumonia (PCP) in AIDS patients.

As many as 80 percent of AIDS patients experience at least one episode of PCP and about one-third of these patients have a recurrence of the disease. Drugs currently used for treatment of acute PCP are toxic to the majority of AIDS patients. The combination of clindamycin and primaquine reduces the numbers of PCP organisms in laboratory tests and in animal studies. Both drugs can be given orally, concentrate in lung tissue, and have been used safely in humans for treatment of other diseases. It is possible that the combination may prove to be as good or better than standard therapy for PCP and side effects may be less.

DETAILED DESCRIPTION:
As many as 80 percent of AIDS patients experience at least one episode of PCP and about one-third of these patients have a recurrence of the disease. Drugs currently used for treatment of acute PCP are toxic to the majority of AIDS patients. The combination of clindamycin and primaquine reduces the numbers of PCP organisms in laboratory tests and in animal studies. Both drugs can be given orally, concentrate in lung tissue, and have been used safely in humans for treatment of other diseases. It is possible that the combination may prove to be as good or better than standard therapy for PCP and side effects may be less.

The proposal for the first 20 patients enrolled in ACTG 044 initially called for an open-labelled, pilot study of intravenous (IV) clindamycin and primaquine therapy in patients with mild to moderate PCP. Preliminary results of the first 22 patients entered into ACTG 044 indicate that the response rate to therapy was over 90 percent. The rate of discontinuation secondary to toxic side effects was only 20 percent. Additional uncontrolled studies have shown an excellent clinical response and safety profile in another 60 patients. The protocol has been amended to provide an all oral dosing regimen. An additional 20 patients with mild PCP will be enrolled and tested with oral clindamycin and primaquine on an outpatient basis. All patients will receive clindamycin and primaquine. Total duration of therapy will be 21 days. Patients may be hospitalized at any time during the study as clinically indicated. Treatment with zidovudine may be started or resumed after completion of clindamycin / primaquine therapy.

AMENDED: An additional 30 patients instead of 20 patients with mild PCP will be enrolled.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Oral antiemetics.

Patients must have the following for inclusion:

* HIV positive by ELISA, p24 antigen or culture.
* Pneumocystis carinii pneumonia (PCP).
* Patients must have an (A-a) DO2 < 40 mmHg on room air.
* Willingness to sign an informed consent.

Prior Medication:

Allowed:

- Prophylaxis for Pneumocystis carinii pneumonia (PCP) with agents other than clindamycin and primaquine.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Hematotoxic therapy, including zidovudine (AZT) or ganciclovir.

Patients with the following are excluded:

* History of allergy to clindamycin, lincomycin, or related drugs; or to primaquine or related drugs.
* Positive screen for G6PD deficiency, known NAD methemoglobin reductase deficiency, and/or known hemoglobin M abnormality.
* Concomitant conditions defined in Patient Exclusion Co-Existing Conditions.
* Any medical or social situation which, in the opinion of the investigator, would adversely affect participation in the study.
* Note:

Patients may be enrolled while G6PD screen is pending, but must be withdrawn if results are not known within 5 days after entry.

Prior Medication:

Excluded within 14 days of study entry:

* Systemic steroids at doses exceeding physiologic replacement or other investigational agents.
* Excluded within 6 weeks of study entry:
* Prior institution of any antiprotozoal therapy for the current episode of Pneumocystis carinii pneumonia or prophylaxis.

Patients must not have any of the following symptoms or diseases:

* History of allergy to clindamycin, lincomycin, or related drugs; or to primaquine or related drugs.
* Positive screen for G6PD deficiency, known NAD methemoglobin reductase deficiency, and/or known hemoglobin M abnormality.
* Diarrhea, defined as = or > 3 watery stools per day.
* Severe nausea and vomiting or other medical condition, such as ileus, that precludes oral therapy.
* Ventilator dependence or (A-a) DO2 = > 30 mm Hg.
* Any medical or social situation which, in the opinion of the investigator, would adversely affect participation in the study.
* Note:

Patients may be enrolled while G6PD screen is pending, but must be withdrawn if results are not known within 5 days after entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Study Completion 1991-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Black JR, Study Chair
Locations (7):
- United States (7):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio

REFERENCES:
- [Background] Black JR, Feinberg J, Murphy RL, Fass RJ, Carey J, Sattler FR. Clindamycin and primaquine as primary treatment for mild and moderately severe Pneumocystis carinii pneumonia in patients with AIDS. Eur J Clin Microbiol Infect Dis. 1991 Mar;10(3):204-7. doi: 10.1007/BF01964465. PMID 2060532
- [Background] Black JR, Feinberg J, Murphy RL, Fass RJ, Finkelstein D, Akil B, Safrin S, Carey JT, Stansell J, Plouffe JF, et al. Clindamycin and primaquine therapy for mild-to-moderate episodes of Pneumocystis carinii pneumonia in patients with AIDS: AIDS Clinical Trials Group 044. Clin Infect Dis. 1994 Jun;18(6):905-13. doi: 10.1093/clinids/18.6.905. PMID 8086551